CLINICAL TRIAL: NCT03542279
Title: Combination Therapy of Pulse Corticosteroid and Plasma Exchange Followed by Intravenous Immunoglobulin in Patients With Severe Antibody- Associated Autoimmune Encephalitis: a Randomized Controlled Trial
Brief Title: CPI Combination Therapy for Autoimmune Encephalitis
Acronym: CPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yan Zhang, Chief physician, professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AE-CPI
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-10

CONDITIONS: Autoimmune Encephalitis
Keywords: Autoimmune encephalitis, Plasma exchange, Immunotherapy, Outcome; corticosteroid; immunoglobulin
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Plasma Exchange; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPI group (Experimental): Intravenous methylprednisolone (IVMP) combined with PE (5 times in each course) and IVIG after PE.
  Interventions: Procedure: Plasma exchange (PE); Drug: intravenous immunmoglobulin (IVIG), intravenous methylprednisolone (IVMP)
- CIP group (Active Comparator): IVMP and IVIG (0.4g/kg/d for 5 days) immediately, followed by PE at least 2 weeks after IVIG treatment.
  Interventions: Procedure: Plasma exchange (PE); Drug: intravenous immunmoglobulin (IVIG), intravenous methylprednisolone (IVMP)

INTERVENTIONS:
Procedure: Plasma exchange (PE) — PE is performed every other day using a multi-filtrate apheresis device (Fresenius, Bad Homburg, Germany), and 5 times in total for each course. The plasma removed during PE is replaced with an equal volume of substitution (half 5% albumin with normal saline and half plasma). The plasma volume to be replaced was estimated according to the following formula: plasma volume (L) = 7.5%×weight (kg)×(1-hematocrit)×1000ml. Heparin was added to the exchange circuit to prevent blood clotting. The exchange rate was monitored, recorded, and balanced to prevent cardiovascular instability. Blood pressure and other vital signs were closely monitored every 15 minutes throughout the exchange.
Drug: intravenous immunmoglobulin (IVIG), intravenous methylprednisolone (IVMP) — IVIG is given 0.4 g/kg/d for each course for 5 days. IVMP is 1,000 mg or 500 mg methylprednisolone for 3 or 5 days, and the dosage of glucocorticoid will gradually decrease.

SUMMARY:
Corticosteroids, intravenous immunoglobulin (IVIG), and plasma exchange (PE) are the first-line therapies for autoimmune encephalitis (AE) patients, but optimal first-line treatment strategy for different AE patients remains undetermined. The study is to compare the efficacy between pulse corticosteroid plus PE initially followed by IVIG (CPI therapy) and pulse corticosteroid plus IVIG followed by PE two weeks later (CIP therapy) in patients with severe antibody-associated autoimmune encephalitis (AE).

DETAILED DESCRIPTION:
Patients with AE will be randomly divided into the CPI and CIP group according to the random table. All patients will receive tumour screening, symptomatic supportive treatment, and immunotherapy. The immunotherapy includes intravenous methylprednisolone (IVMP), intravenous immunoglobulin (IVIG; 0.4 g/kg/d for each course for 5 d), PE and immunosuppressants. Patients in the CPI group received IVMP and PE treatment without delay, followed by IVIG immediately after PE treatment. Patients in the CIP group were given IVMP and IVIG and IVMP immediately, followed by PE at least 2 weeks after IVIG treatment. The patients received long-term immunotherapy involving a combination of oral corticosteroids and immunosuppressants (such as mycophenolate mofetil at a dose of 1-2g/d) for 6-12 months if no contraindications. The primary outcome is the proportion of patients achieving functional improvement [a decrease of at least 1 point in modified Rankin Scale (mRS) score] at 3 months after immunotherapy.

ELIGIBILITY:
Inclusion criteria:

1. 14-65 years old;
2. met all the three following diagnostic criteria of AE: (i) subacute onset (rapid progress of less than 3 months) of working memory deficits, altered mental status, or psychiatric symptoms; (ii) at least one of the followings: new focal CNS findings, seizures not explained by a previously known disease, cerebrospinal fluid (CSF) pleocytosis (white blood cell count 5 cells/mm3), magnetic resonance imaging (MRI) features suggestive of encephalitis, and (iii) reasonable exclusion of alternative causes;
3. the presence of antibody against neuronal surface antigen in serum or CSF indicating a positive diagnosis of AE using a cell-based assay;
4. critically ill with a modified Rankin scale (mRS) score of 4 to 5;
5. within 3 months of onset;
6. no immunotherapy previously.

Exclusion criteria:

1. relative contraindications of TPE treatment: serious underlying diseases such as severe active hemorrhage, disseminated intravascular coagulation, severe hypotension or shock, unstable cardiac failure, cerebral herniation, severe infection or other endangered conditions;
2. allergic to immunoglobulin;
3. contraindications of glucocorticoid therapy: glucocorticoid allergy, active gastric or duodenal ulcer, severe osteoporosis, diabetes, hypertension after recent gastrointestinal anastomosis, and serious infection that cannot be controlled by antibiotics;
4. serious underlying diseases, such as cardiac dysfunction, arrhythmia, and coagulation disorders;
5. premorbid mRS ≥ 3.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
proportion of subjects achieving functional improvement | 3 months following Immunotherapy
  Functional improvement is defined as a decrease of at least 1 point in mRS score, modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.

SECONDARY OUTCOMES:
modified Rankin Scale | 3 months following Immunotherapy
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
modified Rankin Scale | 6 months following Immunotherapy
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
modified Rankin Scale | 12 months following Immunotherapy
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
modified Rankin Scale | 24 months following Immunotherapy
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
proportion of favorable outcome | 3 months following Immunotherapy
  A mRS score of 0-2 was considered a favorable outcome, whereas a mRS score of 3-6 was graded as an unfavorable one.
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
proportion of favorable outcome | 6 months following Immunotherapy
  A mRS score of 0-2 was considered a favorable outcome, whereas a mRS score of 3-6 was graded as an unfavorable one.
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
proportion of favorable outcome | 12 months following Immunotherapy
  A mRS score of 0-2 was considered a favorable outcome, whereas a mRS score of 3-6 was graded as an unfavorable one.
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
proportion of favorable outcome | 24 months following Immunotherapy
  A mRS score of 0-2 was considered a favorable outcome, whereas a mRS score of 3-6 was graded as an unfavorable one.
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
CASE score | 3 months following Immunotherapy
  Clinical Assessment Scale in Autoimmune Encephalitis
CASE score | 6 months following Immunotherapy
  Clinical Assessment Scale in Autoimmune Encephalitis
CASE score | 12 months following Immunotherapy
  Clinical Assessment Scale in Autoimmune Encephalitis
CASE score | 24 months following Immunotherapy
  Clinical Assessment Scale in Autoimmune Encephalitis
Length of ICU stay | before discharge
  Length of ICU stay (days)

OTHER OUTCOMES:
Adverse events | within 24 months following immunotherapy
  Adverse events related with PE

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, MD, Phd, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No